CLINICAL TRIAL: NCT03412656
Title: Assessing the Effectiveness of Upper-limb Force Feedback With the SoftHand Pro Myoelectric Prosthesis in Persons With Transradial Limb Loss
Brief Title: Assessing Force Feedback With the SoftHand Pro
Acronym: CUFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristin Zhao, PhD (Other)
Collaborators: Arizona State University (Other); University of Pisa (Other)
Responsible Party: Sponsor-Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-005611
Record Dates: First submitted 2018-01-21; First posted 2018-01-26 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Amputation, Traumatic; Limb Defect
Keywords: CUFF; Soft Hand Pro; SHP; SH Pro; SoftHand
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Patient (Experimental): Testing will include assessments of activities of daily living (ADLs) by a physical therapist, biomechanical measures of forces applied to objects and motion of the upper limb collected during commonly-performed tasks, and surveys assessing user preference regarding the force feedback feature, all while using the SoftHand Pro myoelectric lower arm prosthetic and the CUFF force feedback devices in tandem, utilizing the subjects' own prosthetic sockets. Grip force will be recorded using sensors attached to the CUFF device. During each session, videos will be obtained of the subjects performing tasks for kinematics analysis. The experimental sessions are organized into one to two sessions, comprising up to 16 hours, as determined by subject availability.
  Interventions: Device: SoftHand Pro with CUFF force feedback device
- Control (Other): Testing will include assessments of activities of daily living (ADLs) by a physical therapist, biomechanical measures of forces applied to objects and motion of the upper limb collected during commonly-performed tasks, and surveys assessing user preference regarding the force feedback feature, all while using the SoftHand Pro myoelectric lower arm prosthetic and the CUFF force feedback devices in tandem, utilizing an adapter simulating a prosthetic socket. Grip force will be recorded using sensors attached to the CUFF device. During each session, videos will be obtained of the subjects performing tasks for kinematics analysis. The experimental sessions are organized into one to two sessions, comprising up to 16 hours, as determined by subject availability.
  Interventions: Device: SoftHand Pro with CUFF force feedback device

INTERVENTIONS:
Device: SoftHand Pro with CUFF force feedback device — Participants will complete various movement and activity of daily living (ADL) assessments to test the effectiveness of the CUFF device in combination with the Soft Hand Pro (SHP) in conveying haptic force feedback to patients with transradial limb loss, and to assess the extent to which the grip force feedback improves the embodiment of the prosthetic device.
  Other Names: SoftHand; SoftHand Pro; CUFF; SHpro

SUMMARY:
The trial is designed to test the effectiveness of a force-feedback cuff in combination with a myoelectric prosthesis in conveying information on grasp strength to the user, as well as the user's preference regarding the feature.

DETAILED DESCRIPTION:
The human sensorimotor control system uses both feedforward planning and sensory feedback information, in order to actuate the musculoskeletal system and interact with the external environment, e.g. when modulating grip force for various object properties. As a result, lack of sensory input, as in the case of motor impairments or amputations, can dramatically affect activities of daily living (ADLs). The contribution of the proposed research will be to test the effectiveness of a novel, non-invasive prosthetic technology in delivering sensory information. The investigators' approach is "modality matching," in that it produces a sensation in the user similar to the type of information to be transmitted. Specifically, the approach will combine the Soft Hand Pro (SHP), an anthropomorphic, myoelectrically controlled prosthetic hand, with an upper limb force feedback device (CUFF) to provide patients with transradial amputations with grasp force (pressure) information.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years.
2. no prior experience with the CUFF device.
3. history of elbow disarticulation, transradial, or transhumeral limb loss (non-control subjects only).

Exclusion Criteria:

1. amputation for less than 6 months
2. clinical history of brachial plexopathy, cervical radiculopathy or polyneuropathy
3. orthopedic, joint degeneration (i.e., arthritis, verified by x-ray) affecting the hand or cervical spine that severely limit upper limb function
4. visual problems that would interfere with the grasp task
5. co-existing central nervous system disease with symptoms that limit upper extremity function (e.g., multiple sclerosis, motor neuron disease, myasthenia gravis, Parkinson's disease, dystonia) revealed in medical history
6. significant rigidity as assessed through range of motion testing
7. active psychiatric illness
8. significant cognitive impairments (a score < 24 on the Mini-Mental State Examination)
9. use of medications that might affect sensory and/or motor functions
10. inability to effectively control myoelectrics for study purposes (control subjects only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Conveyance of force feedback | 1 year
  Assessments will measure the extent to which the CUFF device conveys haptic force feedback, when used in combination with the Soft Hand Pro.
Improvement to device embodiment through addition of grip force feedback | 1 year
  Assessments will determine any improvement of device embodiment from the addition of grip force feedback to the Soft Hand Pro.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin D. Zhao, Ph.D., Principal Investigator — Mayo Clinic; Karen L. Andrews, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials